CLINICAL TRIAL: NCT01508767
Title: Prospective Randomized Controlled Trial of Early Post-operative Removal of Urethral Catheter in Patients Undergoing Colorectal Surgery With Epidural Analgesia
Brief Title: Early Post-operative Removal of Urethral Catheter in Patients Undergoing Colorectal Surgery With Epidural Analgesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College Hospital Galway (Other)
Responsible Party: Principal Investigator, Myles Joyce, Consultant colorectal and general surgeon, University College Hospital Galway
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Joyce-2011
Record Dates: First submitted 2012-01-04; First posted 2012-01-12 (Estimated); Last update posted 2013-08-19 (Estimated); Status verified 2013-08

CONDITIONS: Urinary Retention
MeSH Terms: conditions — Urinary Retention | interventions — Urinary Catheters

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Study group 1 (Experimental): Early removal of urethral catheter 48 hours post-operatively.
  Interventions: Other: Removal of urethral catheter
- Study group 2 (Other): Removal of urethral catheter once epidural analgesia has been withdrawn.
  Interventions: Other: Removal of urethral catheter

INTERVENTIONS:
Other: Removal of urethral catheter — All participants are to have a urethral catheter placed following successful placement of an epidural catheter for analgesia prior to undergoing colorectal resection. Following urethral catheter placement participants will be randomly assigned to either the experimental arm or the control arm. Participants assigned to the experimental arm will have their urethral catheters removed at 48 hours following surgery. Participants assigned to the control group will have their urethral catheters removed within 12 hours of withdrawal of the epidural infusion, as is standard practice in our institution.
  Other Names: Urethral catheter; Indwelling Urinary catheter; Indwelling urethral catheter

SUMMARY:
Patients undergoing colon or rectal surgery will usually have a urinary catheter (silicone tube) placed in the bladder at the time of operating to monitor kidney function during surgery and in the post-surgery period. Such patients will also have an infusion into the spine, known as an epidural, after surgery to provide them with continuous pain relief. Urinary catheters should be removed as early as possible once they are no longer required to facilitate patients becoming mobile after surgery and to reduce the risk of patients developing a urinary tract infection.

Traditionally these catheters are not removed until the patients epidural infusion is withdrawn, as in theory to do so would predispose the patient to developing acute retention of urine due to lack of sensation when the bladder is full. The investigators hypothesis is that urinary catheters placed via the urethra can be withdrawn 48 hours after colon/rectal surgery in patients receiving epidural pain relief without a significant increase in rates of urinary retention.

DETAILED DESCRIPTION:
Patients undergoing colon or rectal surgery will be randomly assigned to one of two groups: Patients in study group 1 (SG1) will have their urinary catheters removed at 48 hours post-operatively; Patients in study group 2 (SG2) will have their urinary catheters removed only after the epidural has been withdrawn in the post-operative period. We will be primarily examining rates of urinary retention in both groups. We will also be examining rates of urinary tract infection, chest infection (frequently a result of poor mobility after surgery), and wound infection and other complications after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18
* Competent to consent to participate in trial
* Undergoing colorectal surgery (any resection of large bowel, formation of colostomy, anterior resection, low anterior resection, panproctocolectomy, abdominoperineal resection).
* Receiving epidural analgesia post-operatively
* If male, international prostate symptom score <20.

Exclusion Criteria:

* Previous lower urinary tract surgery
* Chronic lower urinary tract disease
* Intermittent self-catheterisation
* Neurogenic bladder
* Urethral catheter inserted >24 hours pre-operatively
* Presence of pelvic sepsis/abscess at surgery
* Previous trans-abdominal pelvic surgery
* Urethral catheter required for urine output monitoring beyond 24 hours post-operatively
* Presence of enterovesical fistula
* Pre-operative use of medications which alter detrusor function
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2012-01; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Post-operative urinary retention requiring re-catheterisation | 14 days following urethral catheter removal
  Development of acute post-operative urinary retention demonstrated by a post-void residual >100mls on bladder ultrasound requiring re-catheterisation within 2 weeks of removal of urethral catheter in the post-operative period.

SECONDARY OUTCOMES:
Symptomatic bacteruria | Within 14 days of urethral catheter removal
  Should a patient experience lower urinary tract symptoms following catheter removal a mid-stream urine sample will be taken for microscopy and culture. A pure culture of a single organism of >100,000 colony forming units will be considered a positive culture.
Pulmonary complications | For the first 14 days post-operatively
  The development of post-operative pulmonary complications such as atelectasis, pneumonia occurring within 14 days of surgery will be considered.
Surgical site infection | Within 7 days post-operatively
  The development of wound and other surgical site infections within 7 days of undergoing colorectal surgery will be considered.

CONTACTS AND LOCATIONS:
Overall Officials: Myles R. Joyce, MB, BCh, BAO, Principal Investigator — University College Hospital Galway
Locations (1):
- University College Hospital Galway, Galway, Co. Galway, Ireland

REFERENCES:
- [Derived] Ellahi A, Stewart F, Kidd EA, Griffiths R, Fernandez R, Omar MI. Strategies for the removal of short-term indwelling urethral catheters in adults. Cochrane Database Syst Rev. 2021 Jun 29;6(6):CD004011. doi: 10.1002/14651858.CD004011.pub4. PMID 34184246
- [Derived] Coyle D, Joyce KM, Garvin JT, Regan M, McAnena OJ, Neary PM, Joyce MR. Early post-operative removal of urethral catheter in patients undergoing colorectal surgery with epidural analgesia - a prospective pilot clinical study. Int J Surg. 2015 Apr;16(Pt A):94-98. doi: 10.1016/j.ijsu.2015.03.003. Epub 2015 Mar 10. PMID 25769395